CLINICAL TRIAL: NCT04772521
Title: Evaluation of a Smoking Cessation Program in Workplaces in Hong Kong: a Pragmatic Randomized Controlled Trial on Mobile Phone-Based Intervention on Smoking Cessation and Reducing Mental Health Symptoms
Brief Title: Smoking Cessation Programme in Workplaces in Hong Kong (Phase Ⅴ)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Lok Sin Tong Benevolent Society, Kowloon (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LST SCPW P5
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Personalized chat-based support and nicotine replacement therapy sampling (NRT-S) for continued smokers at 6 months for intervention group
  Interventions: Behavioral: General health talk; Behavioral: Personalized chat-based interactions; Behavioral: Phone follow-up/counselling service; Drug: Mailed nicotine replacement therapy (NRT)
- Control (Placebo Comparator): Regular text-based support and nicotine replacement therapy sampling (NRT-S) for continued smokers at 6 months for control group
  Interventions: Behavioral: General health talk; Behavioral: Text message; Behavioral: Phone follow-up/counselling service; Drug: Mailed nicotine replacement therapy (NRT)

INTERVENTIONS:
Behavioral: General health talk — Health talk provided information about hazards of tobacco (active smoking, second- and third-hand smoke), benefits of quitting smoking and methods to quit smoking.
Behavioral: Personalized chat-based interactions — Individual chat-based interactions last 3 months and consist of 2 parts. First part is regular message. The schedule will be adjusted according to the participants' quitting and mental health status. The second part includes real-time psycho-behavioral intervention delivered by trained cessation counsellors using the acceptance and commitment therapy (ACT) model for smoking cessation and reliving mental health problems. The conversation is based on participants' socio-demographic characteristics, smoking habit at baseline, and updated smoking status and mental health status assessed during online conversation and the baseline questionnaire.
  Arms: Intervention
Behavioral: Text message — Regular messages will be sent twice per month within 3 months. These messages covers simple cessation advice and reminders for follow-ups.
  Arms: Control
Behavioral: Phone follow-up/counselling service — The intervention outcomes and participants' smoking status will be followed up regularly via telephone interviews (15 - 30 minutes).
Drug: Mailed nicotine replacement therapy (NRT) — Full course of NRT treatment (8 weeks) will be provided to all participants who are still smoking at 6-month follow-up and request, or willing to use NRT after advice from counsellors. Medications will be mailed from the smoking cessation clinics.
  Other Names: NRT

SUMMARY:
Smoking causes cardiovascular and respiratory diseases, cancers and diabetes, and it has been a leading risk factor for death globally. Despite the availability of smoking cessation services locally, most smokers do not use such services. Workplace is one of the most convenient platforms to provide smoking cessation services and over 55% of smokers are employed according to the local population-based survey. Moreover, The COVID-19 pandemic and new normal increase in mental health burden to people in the workplace. An online survey during the pandemic found 88% of Hong Kong employees suffered from stress at work during the past 7 days. Mental health can be both precursors and consequences of smoking. However, the effectiveness of a smoking cessation programme conducted in workplace is yet to be examined in Hong Kong, and the mental health support for smoking employees in promoting smoking cessation is not clear. Thus, this study aims to test, by a 2-arm RCT, the effectiveness of an intervention of which includes mobile phone-based intervention on reducing mental health symptoms and smoking cessation in workplaces in Hong Kong; identify facilitators and barriers of successful policy implementation and quitting; examine and evaluate the company environment and their policies in promoting smoking cessation.

DETAILED DESCRIPTION:
This study will separate into two phases. Phase I is a large scale cross-sectional survey of corporations in Hong Kong to examine the employers' knowledge, attitudes and practices in promoting SC in the workplace. Phase II is a 2-arm randomized controlled trial that will be conducted to examine the effectiveness of mobile phone-based intervention combined with company health talk, brief phone counselling and nicotine replacement therapy sampling, for SC in workplaces.

Data analyses

Phase I:

Descriptive statistics will be used to analyze the (1) profile of the corporations, including the total number of employees and smoking employees; (2) employers/managerial staff's knowledge on smoking; (3) employers/managerial staff's attitudes on smoking cessation; (4) practices of the companies with respect to smoking cessation.

Phase II:

Primary outcome is self-reported abstinence in the past 7 days at 6-month follow-up. Secondary outcomes for smoking cessation include self-reported abstinence in the past 7 days at 9- and 12-month follow-ups, the biochemically validated abstinence (defined as exhaled CO level <4ppm and saliva cotinine level ≤30 ng/ml); smoking reduction (50% or above reduction in cigarette consumption compared with baseline. Secondary outcomes for mental health include stress (Perceived Stress Scale-10), depression (Personal Health Questionnaire for Depression), anxiety (Generalized Anxiety Disorder scale) and self-rated health.

Descriptive statistics such as frequency, percentage, and mean will be used to summarize the outcomes and other variables. Chi-square tests and t-tests will be used to compare outcome variables between subgroups. The intention-to-treat (ITT) analysis will be used such that those lost to contact and refused cases at the follow-ups will be treated as no reduction in cigarette consumption nor quitting. Multiple imputations will be used to compute missing data for outcome variables. The association between intervention adherence (e.g., engagement in the IM interaction) and the primary outcome within the participants in the intervention group will be examined. The intervention effect by subgroups will be assessed respectively, including sex, age, education level, company types, previous quit attempts, cigarette dependence, and intention to quit, although the statistical power would be lower due to smaller numbers.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged 18 or above
2. Smoke at least 1 cigarette per day or use e-cigarette (EC) or heated tobacco product (HTP) daily
3. PSS-4 score ≥ 6, or GAD-2 score≥ 3, or PHQ-2 score≥ 3
4. Able to communicate in Cantonese/Mandarin and read Chinese
5. Able to use instant messaging tool (e.g. WhatsApp) for communication.
6. Stay in Hong Kong during the intervention and follow-up periods (12 months)

Exclusion Criteria:

1. Smokers who are psychologically or physically unable to communicate
2. Currently following other smoking cessation program(s)
3. Smokers who have severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Self-reported 7-day point prevalence quit rate | 6-month
  Smokers who did not smoke even a puff in the 7 days preceding the follow-up

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence quit rate | 9-,12-month
  Smokers who did not smoke even a puff in the 7 days preceding the follow-up
Biochemical validation of smoking status | 6-, 9-, and 12-month
  Biochemically validated quit rate (saliva cotinine level and exhale carbon monoxide test)
Self-reported reduction cigarette rate | 6-, 9-, and 12-month
  smoking reduction (50% or above reduction in cigarette consumption compared with baseline).
Self-reported perceived stress | 6-, 9-, and 12-month
  Stress will be assessed by Perceived Stress Scale-4 (PSS-4). It reports perceived stress in the past month on a 5-point Likert scale (0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often, 4 = very often). Individual scores on the PSS can range from 0 to 16 with higher scores indicating higher perceived stress.
Self-reported depression symptoms | 6-, 9-, and 12-month
  Depression will be assessed by Personal Health Questionnaire for Depression-2 (PHQ-2). The PHQ-2 inquires about the frequency of depressed mood and anhedonia over the past two weeks. A PHQ-2 score ranges from 0-6. If the score is 3 or greater, major depressive disorder is likely.
Self-reported anxiety symptoms | 6-, 9-, and 12-month
  Anxiety will be assessed by Generalized Anxiety Disorder-2 (GAD-2). The GAD-2 is a very brief and easy to perform initial screening tool for generalized anxiety. A GAD-2 score ranges from 0-6. If the score is 3 or greater, generalized anxiety disorder is likely.
Self-rated health | 6-, 9-, and 12-month
  Self-rated health will be measured as a single-item with the response items "excellent," "very good," "good," "fair," or "poor."

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No